CLINICAL TRIAL: NCT02848209
Title: Histological Evaluation of Peeling Induced Skin Changes of Different Peeling Agents in Surgically Subcutaneous Undermined Skin Flaps in Facelift Patients
Brief Title: Histological Skin Changes of Different Peeling Agents in Surgically Subcutaneous Undermined Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Ocean Clinic Marbella, Spain (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: PEEL1
Record Dates: First submitted 2016-07-25; First posted 2016-07-28 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2016-07

CONDITIONS: Burn of Face, Head and/or Neck; Peeling
Keywords: Peeling; Histological skin changes; Trichloroacetic acid peel; phenol/croton oil peel
MeSH Terms: interventions — Tooth Exfoliation; Phenol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control (No Intervention): No peeling applied on the skin flap
- Drug: TCA 20% Peeling (Experimental): Trichloroacetic acid 20% applied on the skin flap until even frosting for 2-4 minutes.
  Interventions: Procedure: TCA 20% Peeling
- Drug: TCA 40% Peeling (Experimental): Trichloroacetic acid 40% applied on the skin flap until even frosting for 2-4 minutes.
  Interventions: Procedure: TCA 40% Peeling
- Drug: Phenol/croton oil Peeling (Experimental): Phenol/croton oil applied on the skin flap occluded with silicone tape for 24 hours and not neutralized.
  Interventions: Procedure: Phenol/croton oil Peeling

INTERVENTIONS:
Procedure: TCA 20% Peeling — TCA peel at a concentration of 20% is applied on subcutaneous undermined skin samples for 2 to 4 minutes until even frosting and neutralized at the even frosting Point.
  Arms: Drug: TCA 20% Peeling
Procedure: Phenol/croton oil Peeling — Phenol/croton oil is applied on subcutaneous undermined skin samples and occluded with silicone tape for 24 hours and not neutralized.
  Arms: Drug: Phenol/croton oil Peeling
Procedure: TCA 40% Peeling — TCA peel at a concentration of 40% is applied on subcutaneous undermined skin samples for 2 to 4 minutes until even frosting and neutralized at the even frosting Point.
  Arms: Drug: TCA 40% Peeling

SUMMARY:
The purpose of this study is to examine the histological skin changes induced by different peeling agents (Trichloroacetic acid 25% and 40% and phenol/croton oil) in subcutaneous undermined facial skin flaps.

DETAILED DESCRIPTION:
Written informed consent has to be obtained from 9 random female Caucasian patients aged between 40 and 80 years who will receive a Peeling assisted volume enhancing (PAVE) facelift procedure in Ocean Clinic, Marbella Spain, to take part in the histologic case control study with a within-subjects design.

After completing the facelift, the subcutaneous undermined abundant pre-auricular skin of both sides which is to be resected as consequence of the lift anyhow of each study patient is not resected and split completely in half to yield four samples of the same size, two on each side, without contacting each other in order to prevent any interaction between the peeling agents (n=9 samples per treatment). One sample serves as the control, while the other three samples are each treated with different peeling agents by the same surgeon: Trichloroacetic acid (TCA) peel at concentrations of 20% and 40% and a phenol/croton oil peel. The TCA samples are peeled immediately for 2 to 4 minutes until even frosting and neutralized at the even frosting point. The phenol/croton oil peeled samples are occluded with silicone tape for 24 hours and not neutralized. After 24 hours during the routine in-hospital stay of the patient, the skin samples are resected, the preauricular wound is closed, and all samples are placed in 10 % neutral buffered formalin. The samples are immediately processed, trimmed, embedded, sectioned and stained with haematoxylin and eosin (H&E) by the same researcher. Histological evaluation which will take place in Tuebingen is carried out using a microscope, and pictures are captured at 10x, 25x and 100x magnification using a digital camera. Two trained histological examiners blinded to the study design independently perform histological evaluations. The depth of necrosis in µm is determined by analysing the tissue damage in relation to histological skin layers. All slices are evaluated using light microscopy to assess the mean depth of necrosis in three samples at three different sites for each specimen. The vertical height in µm between the cutaneous basal membrane and the deepest penetration of tissue damage is measured as well as the total thickness of the epidermis and dermis. Based on the histomorphological changes, actual peeling depth is determined and classified analogously to the current classification of burns: superficial, superficial-partial, deep-partial and full thickness.

ELIGIBILITY:
Inclusion Criteria:

* The population consists of all female English-speaking Caucasian patients of the Department for plastic and aesthetic surgery of Ocean Clinic Marbella, Spain, between 40 and 80 years seeking for elective facial rejuvenation with the PAVE-lift technique (peeling assisted volume enhancing Facelift) who give formal written informed consent to take part in the study.

Exclusion Criteria:

* any known cardiac problems like arrhythmia or conduction disorders, such as Wolff Parkinson White Syndrome
* previous facelift surgery
* previous facial peeling
* Fitzpatrick skin type 4, 5 and 6 (dark tanned skin types in which the applied peeling agents are known to lead to unpleasant results such as hypopigmentation and skin lightening)
* any former episode of skin cancer
* any inability to give informed written consent

Ages: 40 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-07; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Peeling depth | 24 hours
  The vertical height in µm between the cutaneous basal membrane and the deepest penetration of tissue damage is measured as well as the total thickness of the epidermis and dermis

SECONDARY OUTCOMES:
Chemical burn grade | 24 hours
  Based on the histomorphological changes, actual peeling depth is determined and classified analogously to the current classification of burns: superficial, superficial-partial, deep-partial and full thickness.

CONTACTS AND LOCATIONS:
Overall Officials: Phillipp Gonser, MD, Principal Investigator — BG Trauma Centre Tuebingen
Locations (1):
- Ocean Clinic, Marbella, Malaga, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kaye KO, Schaller HE, Jaminet P, Gonser P. The PAVE (peeling-assisted volume-enhancing) lift: A retrospective 6-year clinical analysis of a combined approach for facial rejuvenation. J Plast Reconstr Aesthet Surg. 2016 Aug;69(8):1128-33. doi: 10.1016/j.bjps.2016.04.012. Epub 2016 May 4. PMID 27320171
- See also: Homepage of the recruiting and treating clinic — http://www.oceanclinic.net
- See also: Homepage of the evaluating clinic — http://www.bgu-tuebingen.de